CLINICAL TRIAL: NCT03646747
Title: Oxygen Enhanced MRI Measurement in Head and Neck Cancer: Validation and Efficacy of Response.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sally Falk (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor-Investigator, Sally Falk, Research Project Manager, The Christie NHS Foundation Trust
Organization: The Christie NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18_RADIO_133
Record Dates: First submitted 2018-05-03; First posted 2018-08-24 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Head and Neck Cancer
Keywords: head and neck; radiotherapy; magnetic resonance imaging
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Single site, non-randomised basic science study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI scan (Experimental): 10 healthy participants will be asked to undergo two baseline OE-MRI scans with either nasal cannula or facial mask to breathe air and oxygen throughout.
  Following this initial pilot, OE-MRI will be tested in 30 patients with solid head and neck tumours.
  Interventions: Diagnostic Test: MRI scan

INTERVENTIONS:
Diagnostic Test: MRI scan — Additional imaging using MRI scan

SUMMARY:
This is a prospective pilot study to investigate the potential clinical value of oxygen-enhanced magnetic resonance (OE-MRI) biomarkers in head and neck radiotherapy.

DETAILED DESCRIPTION:
This is a prospective pilot study funded by the NIHR. Healthy participants and patients will be recruited in The Christie NHS Foundation Trust and will be asked to undergo oxygen-enhanced magnetic resonance imaging (OE-MRI) and dynamic contrast-enhanced MRI (DCE-MRI). This study builds on the work recently been completed in lung cancer. Clinical data will be collected from patients notes.

Tumour hypoxia is common in solid tumours and associated with poor response to radiotherapy, poor loco-regional control and survival outcomes in head and neck cancer. There is a need to develop non-invasive tests that can measure tumour hypoxia to improve radiotherapy for these patients. The study will involve 3 components:

1. Reproducibility and feasibility: The reproducibility of OE-MRI in head and neck cancer is unknown. Ten healthy participants will be asked to undergo two baseline OE-MRI scans with either nasal cannula or facial mask to breathe air and oxygen throughout. The order of which non-invasive breathing method will be used first will be randomized.

   Following this initial pilot OE-MRI will be tested in 30 patients with solid head and neck tumours. To assess reproducibility in patients 2 OE-MRI will be performed at baseline.
2. Effect of radiotherapy on tumour and normal tissue: OE-MRI and DCE-MRI signals will be measured at baseline before standard radiotherapy treatment begins and at the end of week 2 week and week 4 following the start of radiotherapy. Comparison of hypoxia measurements will be taken.
3. Biological validation: All 30 patients will undergo a diagnostic biopsy as standard of care at their local hospital. Tissue samples will be requested and multi-gene hypoxia signatures will be tested. OE-MRI signals will be compared with tissue sample from the same patient and the presence of changes in tumour known to be associated with hypoxia will be analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or over
2. Able to receive and understand verbal and written information regarding the study and given written informed consent
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
4. Adequate renal function: Calculated creatinine clearance (Cockcroft-Gault) ≥30mL/min
5. Be able to lie comfortably on back for up to 1 hour
6. Be able to tolerate a thermoplastic shell
7. Female patients must meet one of the following criteria:

   i. Postmenopausal for a minimum of one year ii. Surgically sterile iii. Not pregnant, confirmed by B-HCG blood test. iv. Not breastfeeding
8. Cohort A (healthy participants): Up to 10 will be recruited to validate the use of nasal cannula
9. Cohort B (patients): Any patient with HNSCC who is due to start definitive radiotherapy +/- chemotherapy. Up to 30 will be recruited. Each patient prior to recruitment will undergo a diagnostic biopsy at their local hospital as standard of care. The formalin fixed paraffin embedded (FFPE) tumour biopsy sample blocks will be requested from each site and stored in the Manchester Cancer Research Centre (MRCR) and tested for a multi-gene signature.

Exclusion Criteria:

Healthy volunteers or patients with any contraindications to MRI scanning (i.e heart valve replacement, pacemaker, metal implants not approved for MRI, neurostimulators), history of contrast (Gadolinium) allergy or pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of hypoxia in head and neck squamous cell cancer using oxygen enhanced Magnetic resonance imaging (using a range of different MR sequences) | 3 years
  Assessment of hypoxia in head and neck squamous cell cancer using oxygen enhanced Magnetic resonance imaging (using a range of different MR sequences)

SECONDARY OUTCOMES:
Optimal MRI sequence to image participants with head and neck cancer, based on tumour and organ at risk visualisation. | 3 years
  Optimal MRI sequence to image participants with head and neck cancer, based on tumour and organ at risk visualisation.
Treatment response in a number of participants with head and neck cancer treated with radiotherapy +/- systemic therapy | 3 years
  Treatment response in a number of participants with head and neck cancer treated with radiotherapy +/- systemic therapy
Treatment related toxicities in a number of participants with head and neck cancer as assessed during and after treatment completion | 3 years
  Treatment related toxicities in a number of participants with head and neck cancer as assessed during and after treatment completion
Survival outcomes in a number of participants treated with radiotherapy +/- systemic therapy for head and neck cancer | 3 years
  Survival outcomes in a number of participants treated with radiotherapy +/- systemic therapy for head and neck cancer

CONTACTS AND LOCATIONS:
Overall Officials: James O'Connor, Principal Investigator — University of Manchester

IPD SHARING:
Plan to Share IPD: No